CLINICAL TRIAL: NCT01624870
Title: CoreValve Advance-II Study: Best Practices Investigation of Patients Implanted With the Medtronic CoreValve Bioprosthesis.
Brief Title: CoreValve Advance-II Study: Prospective International Post-market Study
Acronym: Advance-II
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: Advance-II
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Aortic Valve Stenosis; Valvular Heart Disease
Keywords: Aortic Valve Stenosis; Valvular Heart Disease; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CoreValve aortic valve: Implantation of CoreValve aortic valve

SUMMARY:
The CoreValve ADVANCE-II Study is a best practices investigation of patients implanted with the Medtronic CoreValve bioprosthesis.

DETAILED DESCRIPTION:
The purpose of the study was to investigate the rate of conduction disturbances after trans-catheter aortic valve implantation of the Medtronic CoreValve device, aiming to characterize best practices. The investigators did not assign study specific interventions to the subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the criteria of labeling indications of the CoreValve System;
* Patient is above the minimum age as required by local regulations to be participating in a clinical trial regardless of gender and race;
* Provided Signed Informed Consent or Data Release Form.

Exclusion Criteria:

* Patients with a device regulating the heart rhythm by pacing (e.g. pacemaker, resynchronization device, implanted defibrillator);
* Patients with a pre-existing class I or class II indication for new pacemaker implantation according to the 2007 ESC guidelines;
* Persistent or permanent atrial fibrillation (except paroxysmal AF);
* Participation in another drug or device study that would jeopardize the appropriate analysis of endpoints of this study.
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic stenosis and at elevated surgical risk are eligible to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sonia Petronio, M.D., Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (9):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Nemocnice Podlesi Trinec, Třinec, Czechia
- Germany (3):
  - Charite, Campus Mitte - Kardiologie Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Heidelberg, Heidelberg
- Italy (2):
  - Istituto Clinico S. Ambrogio, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Erasmus Medical Center Rotterdam, Rotterdam, Netherlands
- Glenfield Hospital Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petronio AS, Sinning JM, Van Mieghem N, Zucchelli G, Nickenig G, Bekeredjian R, Bosmans J, Bedogni F, Branny M, Stangl K, Kovac J, Schiltgen M, Kraus S, de Jaegere P. Optimal Implantation Depth and Adherence to Guidelines on Permanent Pacing to Improve the Results of Transcatheter Aortic Valve Replacement With the Medtronic CoreValve System: The CoreValve Prospective, International, Post-Market ADVANCE-II Study. JACC Cardiovasc Interv. 2015 May;8(6):837-846. doi: 10.1016/j.jcin.2015.02.005. PMID 25999108

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled: All subjects who enrolled in the study
Period: Overall Study
Arm/Group | All Enrolled
Started | 200 (provided informed consent)
Completed | 173 (Completed 6 month follow up)
Not Completed | 27
Not completed — Death | 19
Not completed — Withdrawal by Subject | 1
Not completed — CoreValve not implanted | 6
Not completed — Lost to follow up | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the study
Groups:
- All Enrolled: All subjects enrolled in the study
Arm/Group | All Enrolled
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 95
Region of Enrollment [Number; unit: participants]
  Netherlands | 40
  Czech Republic | 12
  Belgium | 19
  Italy | 51
  United Kingdom | 8
  Germany | 70

OUTCOME MEASURES:

1. Primary Outcome: New-onset Class I or II Indication for Permanent Pacemaker Implantation
Description: The Kaplan-Meier estimate of new-onset class I or II indication for permanent pacemaker implantation at 30 days for implant depth ≤6mm or >6mm. Where class I is defined as evidence and/or general agreement that a given treatment or procedure is beneficial, useful, and effective and class II is defined as conflicting evidence and/or a divergence of opinion about the usefulness/efficacy of a given treatment or procedure according to the 2007 ESC guidelines.
Time Frame: 30 days post procedure
Population: the populations used for this parameter are sub-population of the 194 implanted subjects for whom data of implant depth was available
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- CoreValve Implant Depth ≤6mm: Enrolled subjects implanted with a CoreValve device at an implant depth of ≤6mm
- CoreValve Implant Depth >6mm: Enrolled subjects with a CoreVavle device at an implant depth of >6mm
Arm/Group | CoreValve Implant Depth ≤6mm | CoreValve Implant Depth >6mm
Number analyzed (Participants) | 83 | 109
Percentage of subjects | 13.3 [7.0 to 21.5] | 21.4 [14.1 to 29.6]

2. Secondary Outcome: Combined Safety Endpoint
Description: The Kaplan-Meier estimate of all-cause mortality, major stroke, life threatening (or disabling) bleeding, acute Kidney Injury - Stage 3 (including renal denervation therapy), peri-procedural myocardial infarction or repeat procedure for valve related dysfunction (surgical or interventional). A Kaplan Meier assessment was used to determine the composite rate.
Time Frame: 30 days post procedure
Population: All implanted
Measure: Number; unit: Percentage of subjects
Groups:
- All Implanted: All subjects who were implanted with the CoreValve device. All subjects in whom the procedure was attempted were implanted with the CoreVave device.
Arm/Group | All Implanted
Number analyzed (Participants) | 194
Percentage of subjects | 6.7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 6 months post-implant procedure.
Arm/Group | All Implanted
All-Cause Mortality (participants affected / at risk) | 17/194
Serious Adverse Events (participants affected / at risk) | 113/194
Other Adverse Events (participants affected / at risk) | 151/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Implanted (N=194)
Permanent Pacemaker Implantation (Surgical and medical procedures) | 50 (50)
Stroke-TIA (Vascular disorders) | 9 (9)
Bleeding (Vascular disorders) | 55 (59)
Acute Kidney Injury (Renal and urinary disorders) | 7 (7)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Coronary obstruction (Vascular disorders) | 1 (1)
Vascular access site and access-related complications (Injury, poisoning and procedural complications) | 44 (48)
Valve-related dysfunction requiring repeat procedure (Surgical and medical procedures) | 5 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Implanted (N=194)
Stroke-TIA (Vascular disorders) | 3 (3)
Renal Failure (Renal and urinary disorders) | 7 (7)
Bleeding Event (Vascular disorders) | 31 (32)
Permanent Pacemaker Implantation (Surgical and medical procedures) | 7 (7)
Re-intervention (Surgical and medical procedures) | 1 (1)
Vascular access site and access-related complications (Injury, poisoning and procedural complications) | 29 (29)
Other Adverse Event (General disorders) | 136 (364) — Any other reported adverse event not associated with the use of the study device were collected without a specific adverse event term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less